CLINICAL TRIAL: NCT03913039
Title: Reduction of Prostate Biopsy Morbidity and Hospitalization Through a Modified Biopsy Protocol Bundle and Region-specific Antibiogram
Brief Title: Reduction of Prostate Biopsy Morbidity
Status: Completed | Type: Observational
Sponsor: Maimonides Medical Center (Other)
Responsible Party: Principal Investigator, Ariel Schulman, Principal Investigator, Maimonides Medical Center
Other Study IDs: 2019-03-03
Record Dates: First submitted 2019-04-10; First posted 2019-04-12 (Actual); Last update posted 2022-02-10 (Actual); Status verified 2022-02

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- transperineal protocol: 1. Transperineal biopsy approach with avoidance of rectal flora
  2. MRI-ultrasound fusion-guided biopsies with reduced number of biopsy cores, where clinically indicated
  3. Rectal swab to identify the presence of fluoroquinolone resistant (FQR) bacteria
  4. Multi-antibiotic prophylaxis
  5. Urine culture, prostate tissue culture and rectal swab culture to define contemporary, region-specific antibiotic resistance patterns.
  Interventions: Procedure: Transperineal biopsy Protocol
- Traditional biopsy: 1. Transrectal approach
  2. Standard 12-core template
  3. Surgeon-specific antibiotic prophylaxis
  4. Urine culture, prostate tissue culture and FQR rectal swab culture to define contemporary, region-specific antibiotic resistance patterns.

INTERVENTIONS:
Procedure: Transperineal biopsy Protocol — 1. Transperineal biopsy approach with avoidance of rectal flora
  2. MRI-ultrasound fusion-guided biopsies with reduced number of biopsy cores, where clinically indicated
  3. Rectal swab to identify the presence of fluoroquinolone resistant (FQR) bacteria
  4. Multi-antibiotic prophylaxis
  5. Urine culture, prostate tissue culture and rectal swab culture to define contemporary, region-specific antibiotic resistance patterns.
  Groups: transperineal protocol

SUMMARY:
Prostate biopsy is typically performed via either the transrectal or transperineal approach. This study is a case-control study being done to determine if a novel prostate biopsy protocol incorporating a transperineal approach, rectal swab to detect resistant bacteria and broad antibiotic prophylaxis will reduce infectious complications and hospital readmission compared to current biopsy practices.

DETAILED DESCRIPTION:
This will be a prospective multi-center cohort case-control study comparing a novel transperineal prostate biopsy protocol integrating measures to reduce post procedural infection (Cases) to traditional transrectal prostate biopsies (Controls). Eligible subjects will be identified through administrative records in the Urology clinics affiliated with Maimonides Medical Center. Eligible patients will be counseled about the risks and benefits of participation and offered enrollment into the study. Demographic data including age, comorbidities and past medical history will be extracted from the medical record.

Men meeting inclusion/exclusion criteria will be prospectively enrolled. The novel transperineal protocol will include the following: (Cases)

1. Transperineal biopsy approach with avoidance of rectal flora
2. MRI-ultrasound fusion-guided biopsies with reduced number of biopsy cores, where clinically indicated
3. Rectal swab to identify the presence of fluoroquinolone resistant (FQR) bacteria
4. Multi-antibiotic prophylaxis
5. Urine culture, prostate tissue culture and rectal swab culture to define contemporary, region-specific antibiotic resistance patterns.

Traditional biopsy protocol includes: (Controls)

1. Transrectal approach
2. Standard 12-core template
3. Surgeon-specific antibiotic prophylaxis
4. Urine culture, prostate tissue culture and FQR rectal swab culture to define contemporary, region-specific antibiotic resistance patterns.

ELIGIBILITY:
Inclusion Criteria:

* Male patients greater than 18 years of age
* Indication for prostate biopsy

Exclusion Criteria:

* Female patients
* Male patients under 18 years of age
* No indication for prostate biopsy

Ages: 18 Years to 120 Years | Sex: Male
Age Groups: Adult, Older Adult
Gender Based: Yes — Assessment of Prostate Cancer treatment - - only males qualify.
Study Population: Males with clinical indication for a prostate biopsy.
Sampling Method: Non-Probability Sample
Enrollment: 157 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Rate of clinically significant post-biopsy complications | 30 Days
  1. Rate of any clinically significant post-biopsy complications including infectious complications and hospital readmissions within 30 days.

SECONDARY OUTCOMES:
1. Number of individual complications within 30 days | 30 Days
  1. Individual complications within 30 days including urinary retention, hematuria, urinary tract infection, hospitalization

CONTACTS AND LOCATIONS:
Locations (1):
- Maimonides Medical Center, Brooklyn, New York, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-04): https://cdn.clinicaltrials.gov/large-docs/39/NCT03913039/Prot_SAP_000.pdf